CLINICAL TRIAL: NCT06410417
Title: The Effect of Reducing Ejaculation Abstinence Time on Assisted Reproductive Technology Outcomes: a Prospective Randomized Controlled Study
Brief Title: Ejaculation Abstinence Time and Assisted Reproductive Technology Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HS-035
Record Dates: First submitted 2024-04-25; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-04

CONDITIONS: Fertilization in Vitro
Keywords: in vitro fertilization; intracytoplasmic sperm injection; Abstinence time; Clinical pregnancy rate; Embryo quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short abstinence time group (Experimental): abstinence time is less than 48 hours
  Interventions: Behavioral: Shorten abstinence time
- routine abstinence time group (No Intervention): Abstinence for 3-7 days

INTERVENTIONS:
Behavioral: Shorten abstinence time — In the experimental group, male ejaculates once on human chorionic gonadotropin trigger day, and can be ejaculated on the second day if ejaculates fail.
  Arms: Short abstinence time group

SUMMARY:
The goal of this clinical trial is to learn if reducing the ejaculation abstinence time can improve the outcome of assisted reproductive technology. The main questions it aims to answer are:

Does reducing the duration of ejaculation abstinence improve the clinical pregnancy rate for in vitro fertilization and intracytoplasmic sperm injection? Does reducing the duration of ejaculation abstinence improve embryo quality in in vitro fertilization and intracytoplasmic sperm injection？ Does reducing the duration of ejaculation abstinence affect pregnancy loss and live birth rates in in vitro fertilization and intracytoplasmic sperm injection?

Researchers will compare less than 48 hours of abstinence time to more than 48 hours, to see if less than 48 hours of abstinence time improved in vitro fertilization outcomes

Participants will:

Control group abstinence for 3-7 days

The experimental group ejaculated once on human chorionic gonadotropin trigger day

Follow up their in vitro fertilization outcomes

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if reducing the ejaculation abstinence time can improve the outcome of assisted reproductive technology.

Group A: Experimental group: ejaculation once within 48 hours before the day of egg retrieval.

Group B: Control group: ejaculation once within 4-7 days before the day of egg retrieval.

There is currently no clear abstinence period for in vitro fertilization, and the usual practice is to refer to the World Health Organization standard for semen testing: abstinence period of 2-7 days.Group A ejaculated once 48 hours before egg retrieval.Group B was the control group, and ejaculation was performed according to the conventional protocol.Most IVF intervals from ovulation initiation to human chorionic gonadotropin trigger day range from 8-11 days, but the fixed time of egg retrieval is 34-37 hours after the trigger day.Therefore, when determining the human chorionic gonadotropin time, it is less than 48 hours before egg retrieval.In the experimental group, male ejaculates once on the trigger day, and can be ejaculated on the second day if ejaculates fail.

Follow up their in vitro fertilization outcomes

ELIGIBILITY:
Inclusion Criteria:

* The couple is between 20 and 45 years old, and the woman's body mass index is greater than 18.5 and less than 30kg/m2.
* Meet the indications of assisted reproductive technology, agree to use assisted reproductive technology to assist pregnancy and have entered the process.
* The male has normal ejaculation function and plans to provide a semen sample by masturbation method on the day of egg retrieval.

Exclusion Criteria:

* Couples with serious infections and major physical diseases, such as HIV.
* The use of testicular sperm for intracytoplasmic sperm injection, such as the azoospermia.
* The use of frozen sperm for assisted reproductive technology.
* Endometriosis, repeated implantation failure, etc.
* There are clear factors affecting semen parameters within 3 months before sperm extraction, including high temperature, contact with chemicals，radiation or drugs that affect sperm, etc.;Previous orchitis/epididymitis, cryptorchidism, receiving radiotherapy and chemotherapy treatment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The pregnancy rate of different abstinence periods in in vitro fertilization. | A year
  All participants underwent ultrasound examination four weeks after embryo transfer. A gestational sac was considered a clinical pregnancy (+), while the absence of a gestational sac was considered a non-clinical pregnancy (-).
  Clinical pregnancy rate = (number of clinical pregnancy (+) cycles/transplant cycles) ×100%.
  The aim was to compare the difference in pregnancy rates between the two groups.
The fertilization rate of different abstinence periods in in vitro fertilization. | A year
  Fertilization rate = (number of fertilized eggs/number of eggs harvested) ×100%.
  The above parameters were evaluated by experienced embryologists according to the evaluation criteria and recorded in the medical record.
  The aim was to compare the difference in fertilization rate between the two groups.
The high-quality embryo rate of different abstinence periods in in vitro fertilization. | A year
  High-quality embryo rate = (number of high-quality embryos/number of normal fertilized cleavage embryos) ×100%.
  The above parameters were evaluated by experienced embryologists according to the evaluation criteria and recorded in the medical record.
  The aim was to compare the difference in high-quality embryo rate between the two groups.

SECONDARY OUTCOMES:
The pregnancy loss rate of different abstinence periods in in vitro fertilization. | 1.5 years
  Pregnancy loss rate = number of pregnancy loss cycles/transplant cycles ×100%. Follow-up should be conducted for couples who are already clinically pregnant to record any pregnancy loss that occurs within 24 weeks of gestation.
  The aim was to compare the difference in pregnancy loss rate between the two groups.
The live birth rates of different abstinence periods in in vitro fertilization. | 1.5 years
  Live birth rate = number of live birth cycles/transplant cycles ×100%. Translation: Continued follow-up is advised for couples who are already clinically pregnant to document the number of live births.
  The aim was to compare the difference in live birth rates between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yueying Zhu, Master, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Result] Vander Borght M, Wyns C. Fertility and infertility: Definition and epidemiology. Clin Biochem. 2018 Dec;62:2-10. doi: 10.1016/j.clinbiochem.2018.03.012. Epub 2018 Mar 16. PMID 29555319
- [Result] Agarwal A, Mulgund A, Hamada A, Chyatte MR. A unique view on male infertility around the globe. Reprod Biol Endocrinol. 2015 Apr 26;13:37. doi: 10.1186/s12958-015-0032-1. PMID 25928197
- [Result] Cates W, Farley TM, Rowe PJ. Worldwide patterns of infertility: is Africa different? Lancet. 1985 Sep 14;2(8455):596-8. doi: 10.1016/s0140-6736(85)90594-x. PMID 2863605
- [Result] Barbagallo F, Condorelli RA, Mongioi LM, Cannarella R, Cimino L, Magagnini MC, Crafa A, La Vignera S, Calogero AE. Molecular Mechanisms Underlying the Relationship between Obesity and Male Infertility. Metabolites. 2021 Dec 4;11(12):840. doi: 10.3390/metabo11120840. PMID 34940598
- [Result] Barbagallo F, Condorelli RA, Mongioi LM, Cannarella R, Aversa A, Calogero AE, La Vignera S. Effects of Bisphenols on Testicular Steroidogenesis. Front Endocrinol (Lausanne). 2020 Jun 30;11:373. doi: 10.3389/fendo.2020.00373. eCollection 2020. PMID 32714277
- [Result] Leisegang K, Dutta S. Do lifestyle practices impede male fertility? Andrologia. 2021 Feb;53(1):e13595. doi: 10.1111/and.13595. Epub 2020 Apr 24. PMID 32330362
- [Result] Fedder J. Nonsperm cells in human semen: with special reference to seminal leukocytes and their possible influence on fertility. Arch Androl. 1996 Jan-Feb;36(1):41-65. doi: 10.3109/01485019608987883. PMID 8824667
- [Result] Gervasi MG, Visconti PE. Molecular changes and signaling events occurring in spermatozoa during epididymal maturation. Andrology. 2017 Mar;5(2):204-218. doi: 10.1111/andr.12320. PMID 28297559
- [Result] Agarwal A, Saleh RA, Bedaiwy MA. Role of reactive oxygen species in the pathophysiology of human reproduction. Fertil Steril. 2003 Apr;79(4):829-43. doi: 10.1016/s0015-0282(02)04948-8. PMID 12749418
- [Result] Zini A, Boman JM, Belzile E, Ciampi A. Sperm DNA damage is associated with an increased risk of pregnancy loss after IVF and ICSI: systematic review and meta-analysis. Hum Reprod. 2008 Dec;23(12):2663-8. doi: 10.1093/humrep/den321. Epub 2008 Aug 29. PMID 18757447
- [Result] Osman A, Alsomait H, Seshadri S, El-Toukhy T, Khalaf Y. The effect of sperm DNA fragmentation on live birth rate after IVF or ICSI: a systematic review and meta-analysis. Reprod Biomed Online. 2015 Feb;30(2):120-7. doi: 10.1016/j.rbmo.2014.10.018. Epub 2014 Nov 13. PMID 25530036
- [Result] Gil-Guzman E, Ollero M, Lopez MC, Sharma RK, Alvarez JG, Thomas AJ Jr, Agarwal A. Differential production of reactive oxygen species by subsets of human spermatozoa at different stages of maturation. Hum Reprod. 2001 Sep;16(9):1922-30. doi: 10.1093/humrep/16.9.1922. PMID 11527899
- [Result] Sorensen F, Melsen LM, Fedder J, Soltanizadeh S. The Influence of Male Ejaculatory Abstinence Time on Pregnancy Rate, Live Birth Rate and DNA Fragmentation: A Systematic Review. J Clin Med. 2023 Mar 13;12(6):2219. doi: 10.3390/jcm12062219. PMID 36983220
- [Result] Chen GX, Li HY, Lin YH, Huang ZQ, Huang PY, Da LC, Shi H, Yang L, Feng YB, Zheng BH. The effect of age and abstinence time on semen quality: a retrospective study. Asian J Androl. 2022 Jan-Feb;24(1):73-77. doi: 10.4103/aja202165. PMID 34747722
- [Result] Agarwal A, Gupta S, Du Plessis S, Sharma R, Esteves SC, Cirenza C, Eliwa J, Al-Najjar W, Kumaresan D, Haroun N, Philby S, Sabanegh E. Abstinence Time and Its Impact on Basic and Advanced Semen Parameters. Urology. 2016 Aug;94:102-10. doi: 10.1016/j.urology.2016.03.059. Epub 2016 May 16. PMID 27196032
- [Result] Gupta S, Singh VJ, Fauzdar A, Prasad K, Srivastava A, Sharma K. Short Ejaculatory Abstinence in Normozoospermic Men is Associated with Higher Clinical Pregnancy Rates in Sub-fertile Couples Undergoing Intra-Cytoplasmic Sperm Injection in Assisted Reproductive Technology: A Retrospective Analysis of 1691 Cycles. J Hum Reprod Sci. 2021 Jul-Sep;14(3):273-280. doi: 10.4103/jhrs.jhrs_235_20. Epub 2021 Sep 28. PMID 34759617
- [Result] Periyasamy AJ, Mahasampath G, Karthikeyan M, Mangalaraj AM, Kunjummen AT, Kamath MS. Does duration of abstinence affect the live-birth rate after assisted reproductive technology? A retrospective analysis of 1,030 cycles. Fertil Steril. 2017 Dec;108(6):988-992. doi: 10.1016/j.fertnstert.2017.08.034. Epub 2017 Oct 31. PMID 29100624
- [Result] Sanchez-Martin P, Sanchez-Martin F, Gonzalez-Martinez M, Gosalvez J. Increased pregnancy after reduced male abstinence. Syst Biol Reprod Med. 2013 Oct;59(5):256-60. doi: 10.3109/19396368.2013.790919. Epub 2013 May 8. PMID 23651301